CLINICAL TRIAL: NCT04350671
Title: An Investigation Into Beneficial Effects of Interferon Beta 1a, Compared to The Base Therapeutic Regiment in Moderate to Severe COVID-19: A Randomized, Double-Blind, Placebo-Controlled, Clinical Trial
Brief Title: Interferon Beta 1a in Hospitalized COVID-19 Patients
Acronym: IB1aIC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Seyed Sina Naghibi Irvani, MD, MPH, MBA, Senior Researcher., Dr., Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Interferon Beta 1a in COVID-19
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: COVID-19; Novel Coronavirus; Interferon Beta 1a; Lopinavir/Ritonavir; Kaletra; Chloroquine; Hydroxychloroquine; Interferon; SARS-CoV-2; 2019-nCoV
MeSH Terms: conditions — COVID-19 | interventions — Interferon beta-1a; Lopinavir; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: The present study is a randomized, double-blind, placebo-controlled, clinical trial, with the approval of the ethics committee will be conducted on patients who have a positive test confirming COVID-19 in Loghman Hakim Medical Education Center in Tehran. Patients will be randomly assigned to the two arms of the study and after completing the course of treatment and collecting and analyzing the necessary information from each patient, the results of the study will be published both on this site and in the form of an article in a reputable international journal.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interferon-β 1a (Experimental): Interferon-β 1a + Lopinavir / Ritonavir + Single Dose of Hydroxychloroquine
  Interventions: Drug: Interferon Beta-1A; Drug: Lopinavir / Ritonavir; Drug: Single Dose of Hydroxychloroquine
- Control (Active Comparator): Lopinavir / Ritonavir + Single Dose of Hydroxychloroquine
  Interventions: Drug: Lopinavir / Ritonavir; Drug: Single Dose of Hydroxychloroquine

INTERVENTIONS:
Drug: Interferon Beta-1A — This will be drug only used in the intervention arm of our study, designed mainly to assess the additional efficacy and safety of Interferon-β 1a in COVID-19 patients.
  Arms: Interferon-β 1a
Drug: Lopinavir / Ritonavir — This Drug will be used in all arms as mandated by our governmental guidelines.
Drug: Single Dose of Hydroxychloroquine — This Drug will be used in all arms as mandated by our governmental guidelines.

SUMMARY:
The present study is a randomized, double-blind, placebo-controlled, clinical trial, with the approval of the ethics committee will be conducted on patients who have a positive test confirming COVID-19 in Loghman Hakim Medical Education Center in Tehran. Patients will be randomly assigned to the two arms of the study and after completing the course of treatment and collecting and analyzing the necessary information from each patient, the results of the study will be published both on this site and in the form of an article in a reputable international journal.

DETAILED DESCRIPTION:
According to previous studies, IFN-β, amongst IFN-1s, has strong antiviral activity and also has an acceptable safety profile. Based on possible therapeutic effects, We decided to lead An Investigation into Beneficial Effects of Interferon Beta 1a, Compared to Interferon Beta 1b And The Base Therapeutic Regiment in Moderate to Severe COVID-19. In a 2003 study, SARS was treated with different human interferons and found that IFN-β was 5 to 10 times more effective than other types of interferons and the strongest antiviral drug possible against SARS-CoV.

Chloroquine has been a broadly-utilized anti-malaria agent which back in 2006, had been proved to be a powerful wide-spectrum antiviral. Moreover, Chloroquine has the characteristics of anti-inflammatory and immune-modulatory by inhibiting the production of TNF-α along with IL-6. In the first half of February, Wang et al illustrated puissant inhibition of SARS-CoV-2 by Chloroquine, when taking two 500-mg tablets of it by mouth per day; similar to some clinical studies in China through this outbreak. According to the news briefing of works of Per Gao et al., it was indicated that chloroquine phosphate actually outdo the control treatment in inhibition of pneumonia exacerbation, improving lung imaging findings, and curtailing the disease course. X. Yao et al. evaluated the possible doses of CQ and HCQ to find the optimized dose in treatment of COVID-19. They revealed that while within in-vitro settings Hydroxychloroquine is more potent than chloroquine. As a conclusion, they suggested a 800 mg daily dose of hydroxychloroquine, followed by an overall maintenance dose of 400 mg per day divided in two separate doses, which was three-fold more potent compared to the 500 mg twice daily administration of chloroquine in 5 days. The new study of Gautret et al. published in 16th March, pointed out that hydroxychloroquine was notably effectual in eradicating SARS-CoV-2 from the nasopharynx. Currently the evidence is quite inconclusive about the effectiveness or comparative effectiveness of either HCQ or CQ. Moreover, CQ has recently become scarce and even unavailable for ordering due to a huge demand for it, all because of a significant interest gained as a potential medicinal alternative for the management of COVID-19. In spite of all, the primary experience in China and France is propitious for the potential role of chloroquine, or alternatively hydroxychloroquine, for managing COVID-19.

Lopinavir, classified in the drug group of protease inhibitors, is utilized for the treatment of patients affected prolongedly with HIV-1. The mechanism by which Lopinavir acts is blocking the main protease of SARS-CoV-1, resulting in inhibition of viral replication. Real-world information supporting the treatment of COVID-19 with LPV/r keep coming out. Chu et al. have discovered that LPV/r has an anti-SARS-CoV effect within both in-vitro settings and clinical studies. In disclosed results of Young and colleagues' research on COVID-19 patients in Singapore, 5 cases received LPV/r monotherapy. Among those 5 patients, 3 had decrease in oxygen requirements after treatment, while the other 2 had their conditions worsened to the point of respiratory failure. Other published evaluations from Korea and China made up of a total of 6 patients, show reduced viral load, and clinical improvement after onset of LPV/r treatment. Latterly, Cao and colleagues illustrated the results of comparing twice a day use of LPV/r 400/100 mg to standard care, for treating the pneumonia caused by SARS-CoV-2. This study's upshot, demonstrated no benefit regarding a lopinavir-ritonavir treatment beyond standard care. Considering the currently available data, it is yet to be determined whether LPV/r could significantly affect the status of COVID-19 patients, either as monotherapy or in combination-therapy. Moreover, close monitoring is needed during the administration of this drug, because particularly elevated levels of AST or ALT suggesting the gastrointestinal complications and hepatoxicity may exclude patients with COVID-19 from clinical trials.

The present study is a randomized, double-blind, placebo-controlled, clinical trial, with the approval of the ethics committee will be conducted on patients who have a positive test confirming COVID-19 in Loghman Hakim Medical Education Center in Tehran. Patients will be randomly assigned to the two arms of the study and after completing the course of treatment and collecting and analyzing the necessary information from each patient, the results of the study will be published both on this site and in the form of an article in a reputable international journal.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50
* COVID-19 Confirmed Cases (Either RT-PCR or CT Scan Confirmed).
* Tympanic Temperature of ≥37.5 AND at least one of the following: Cough, Sputum production, nasal discharge, myalgia, headache or fatigue) on admission.
* Time of onset of the symptoms should be acute ( Days ≤ 10).
* SpO2 ≤ 88%
* Respiratory Rate ≥ 24

Exclusion Criteria:

* Refusal to participate expressed by patient or legally authorized representative if they are present.
* Patients with prolonged QT or PR intervals, Second or Third Degree heart block, Arrhythmias including torsade de pointes
* Patients using drugs with potential interaction with Umifenovir Hydroxychloroquine, Lopinavir/Ritonavir or Interferon-β 1a.
* Pregnant or lactating women.
* History of alcohol or drug addiction in the past 5 years.
* Blood ALT/AST levels > 5 times the upper limit of normal on laboratory results.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2020-04-20 (Estimated); Study Completion 2020-04-24 (Estimated)

PRIMARY OUTCOMES:
Time to clinical improvement | From date of randomization until 14 days later.
  Improvement of two points on a seven-category ordinal scale (recommended by the World Health Organization: Coronavirus disease (COVID-2019) R&D. Geneva: World Health Organization) or discharge from the hospital, whichever came first.

SECONDARY OUTCOMES:
Mortality | From date of randomization until 14 days later.
  If the patient dies, we have reached an outcome.
SpO2 Improvement | Days 1, 2, 3, 4, 5, 6, 7 and 14
  Pulse-oxymetry
Incidence of new mechanical ventilation use | From date of randomization until 14 days later
  Incidence of new mechanical ventilation use
Duration of hospitalization | From date of randomization until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 14 days.
  Duration of hospitalization (days)
Cumulative incidence of serious adverse events | Days 1, 2, 3, 4, 5, 6, 7 and 14.
  With incidence of any serious adverse effects, the outcome has happened.

CONTACTS AND LOCATIONS:
Overall Officials: Ilad Alavi Darazam, MD, Study Chair — Shahid Beheshti University of Medical Sciences; Shervin Shokouhi, MD, Study Director — Shahid Beheshti University of Medical Sciences; Minoosh Shabani, MD, Principal Investigator — Shahid Beheshti University of Medical Sciences; Mohammadreza Haji Esmaelie, MD, Principal Investigator — Shahid Beheshti University of Medical Sciences; Seyed Sina Naghibi Irvani, MD, MPH, MBA, Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- Loghman Hakim Hospital, Shahid Beheshti University of Medical Sciences and Health Services, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided
There is no further information.